CLINICAL TRIAL: NCT04074252
Title: Coupling the Surveillance of Mobility Impaired Adults With Large-Scale Assistive Device Donations and the Suitability of the Long-Term Use of Lofstrand (Forearm) Versus Axillary (Underarm) Crutches Among Mobility Impaired Adults in the Northern Region of Malawi
Brief Title: Mobility Impairment in the Northern Region of Malawi
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to complete intervention due to logistics.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Project Malawi (Unknown)
Responsible Party: Principal Investigator, Rachel Thompson, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-000773
Record Dates: First submitted 2019-06-10; First posted 2019-08-30 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lofstrand Crutches (Active Comparator): This group is given a set of Lofstrand crutches.
  Interventions: Device: Lofstrand Crutches
- Axillary Crutches (Active Comparator): This group is given a set of axillary crutches.
  Interventions: Device: Axillary Crutches

INTERVENTIONS:
Device: Lofstrand Crutches — Device: Set of Lofstrand Crutches
  Arms: Lofstrand Crutches
Device: Axillary Crutches — Device: Set of Axillary Crutches
  Arms: Axillary Crutches

SUMMARY:
The purpose of this study is to investigate whether Lofstrand or axillary crutches are better suited to treat mobility impairments and improve physical activity levels in rural, resource-limited, settings like the Northern Region of Malawi. To do this, we are proposing the implementation of a randomized controlled trial (RCT) to measure and compare the physical activity and satisfaction of mobility aid recipients sorted into two groups - one receiving a set of Lofstrand crutches (Group 1) and the other a set of axillary crutches (Group 2). Changes in physical activity, disability, and life satisfaction levels will measured with a follow-up data collection period conducted one year after the distribution of the devices.

DETAILED DESCRIPTION:
STAGE 1 - BASELINE DATA COLLECTION:

* Potential participants will be identified at outreach clinics in the Mzimba, Rumphi, and Nkhata Bay Districts for participation in the study.
* Potential participants will take the Washington Group Extended Set Questions on Disability (WGES) and those that meet a baseline level of disability/mobility impairment - validated by physiotherapist opinion - are invited to participate in the study.
* 100 or more participants (50+ per group) who fulfill the inclusion criteria will be selected for participation.
* Participants will complete a Demographic Survey to determine their age, gender, health barriers, social determinants of health etc.
* Participants will complete the Global Physical Activity Questionnaire (GPAQ) to determine a baseline of their physical activity.
* Participants will complete the PROMIS Satisfaction with Participation in Social Roles - Short Form 8a (SPSR) and General Life Satisfaction (Ages 18+) - Fixed Form A (GLS) questionnaires to determine a baseline of their overall life satisfaction.
* Treatment groups will be randomized through the use of randomization envelopes.
* Selected devices, as determined in the randomization process, will be distributed to participants in each treatment group.
* The addresses/villages of residences of selected participants will be recorded and marked manually on a detailed satellite map. A list of study participants will be provided to the local Health Surveillance Assistant (HSA) for record keeping and monitoring purposes. (HSAs have intimate knowledge of the communities they serve and will be useful partners to help find participants in the follow-up stages of the trial.)

STAGE 2 - ONE-YEAR FOLLOW-UP DATA COLLECTION:

* Participants will be located using the assistance of the local HSA, address records, and map markings from Stage 1.
* Participants will complete follow-up SPSR, GLS, WGES and GPAQ questionnaires, and will complete the Crutch Satisfaction Survey.
* Reports of missing and damaged crutches will be taken.

STAGE 3 - DATA ANALYSIS:

The two study groups will be compared using the following metrics:

* Stratified by level of disability based on Washington Group Extended Set Questions on Disability
* Changes in GLS and SPSR scores between baseline and follow-up data collection will be used to determine changes in participants' overall life satisfaction.
* Changes in Global Physical Activity Questionnaire scores between baseline and follow-up data collection will be used to determine changes in participants' mobility impairments and day-to-day activity levels.
* Scores from the Crutch Satisfaction Survey will be used determine participants' subjective experiences with their respective mobility devices.

ELIGIBILITY:
Inclusion Criteria:

* Persons fluent in English, Tumbuka, and/or Chichewa.
* Persons diagnosed with a moderate to severe mobility impairment and/or lower extremity disabilities as determined by the WGES Questions on Disability.
* Persons untreated or undertreated for mobility impairment. We consider undertreated persons as those treating their mobility impairments with self-made devices (i.e. wooden crutches or walking sticks), or with devices considered lower than standard of care for their level of impairment (i.e. using a cane instead of crutches).
* Persons who are candidates for both axillary and Lofstrand crutch treatment - as determined by gait analysis conducted by local physiotherapists.
* Persons accessing one of the following 15 outreach distribution clinics located throughout the Mzimba, Rumphi, and Nkhata Bay Districts: Mzuzu Central Hospital, Ekwendeni Mission Hospital, Mtwalo Health Centre, Rumphi MAP Office, Bolero Health Centre, Hewe Health Centre, Livingstonia Mission Hospital, Mhuju Health Centre, Mzimba District Hospital, Jenda Health Centre, Nkhata Bay District Hospital, Mpamba Health Centre, Maula Health Centre, Chintheche Health Centre, and Kande Health Centre.

Exclusion Criteria:

* Persons diagnosed with degenerative conditions that may lead to further deterioration in mobility between data collection periods (i.e. ALS, Muscular Dystrophy, Corticobasal Degeneration etc.)
* Persons with developmental delays that will preclude them from participation in any of the surveys
* Persons with upper extremity disabilities that may preclude them from using crutches.
* Persons who are not permanent residents of the area or have any plans on moving out of the area.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change in scores between baseline and follow-up from the Global Physical Activity Questionnaire (QPAQ) | Baseline and 1 year
  Questionnaire used to measure the patient's self reported level of physical activity. There are 16 questions total. The majority of the questions are binary, but there are a few questions that include a measurement of time (in minutes, hours, and days). There is a numerical output.

SECONDARY OUTCOMES:
Change in scores between baseline and follow-up from the PROMIS Satisfaction with Participation in Social Roles (SPSR) survey | Baseline and 1 year
  Questionnaire used to measure the patient's self reported level of satisfaction with current social roles. There are 7 ordinal type questions, each with 5 different rating options to choose from. There is a numerical output.
Change in scores between baseline and follow-up from the PROMIS General Life Satisfaction (GLS) survey | Baseline and 1 year
  Questionnaire used to measure the patient's self reported level of satisfaction with general life satisfaction. There are 7 ordinal type questions, each with 5 different rating options to choose from. There is a numerical output.
Satisfaction Survey | 1 year
  Questionnaire used to measure the patient's self reported satisfaction with their assigned devices. There is a numerical output.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel M Thompson, MD, Principal Investigator — UCLA/OIC
Locations (1):
- Orthopaedic Institute for Children, Los Angeles, California, United States